CLINICAL TRIAL: NCT00464126
Title: The Use of Colloid Versus Crystalloid in Post-operative Pediatric Cardiac Patients for Fluid Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#: 020775
Record Dates: First submitted 2006-08-18; First posted 2007-04-20 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Diseases
Keywords: crystalloid; colloid; pediatric; cardiac; resuscitation; Postoperative
MeSH Terms: conditions — Heart Diseases | interventions — Albumins; Colloids; Crystalloid Solutions; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colloid (Active Comparator): 5% albumin for volume resuscitation
  Interventions: Other: 5% albumin
- Crystalloid (Placebo Comparator): Saline for volume resuscitation
  Interventions: Other: crystalloid

INTERVENTIONS:
Other: 5% albumin — 5% albumin in 10cc/kg aliquots for postoperative volume resuscitation
  Other Names: colloid; albumin
  Arms: Colloid
Other: crystalloid — saline in 10cc/kg aliquots for postoperative volume resuscitation
  Other Names: saline
  Arms: Crystalloid

SUMMARY:
The purpose of the study is to help determine if either crystalloid solution or colloid solution is more advantageous as a resuscitative fluid in post-operative pediatric cardiac patients.

DETAILED DESCRIPTION:
The study is designed to help detect if there is an advantage in giving one type of resuscitative fluid versus another in the setting of post-operative pediatric cardiac patients. The two types of fluid being compared are crystalloid solution (normal saline) and colloid solution (5% albumin). The primary outcome measurement will be how much volume of each type of fluid will be required in order to maintain hemodynamic stability as determined by mean arterial blood pressure within predetermined parameters. Other secondary outcomes will include determinations of lactate clearance, inotropic support requirements, urine output, peripheral and pulmonary edema that occurs post-operatively, and the over all costs for each fluid based on number of required boluses and number of hours on mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart defect with two ventricle anatomy and physiology
* Ages: 0 - 36 months of age

Exclusion Criteria:

* History of bleeding disorder
* History of renal disorder

Ages: 1 Day to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
maintenance of hemodynamic stability according to an age specific, predetermined, minimal mean arterial blood pressure | Throughout the post operative period

SECONDARY OUTCOMES:
lactate clearance | Throughout the post operative period
inotropic requirements | throughout the post operative period
establishment of adequate urine output | Throughout the post operative period
post-operative occurrence of edema (peripheral and pulmonary) | Througout the post operative period
monitoring of cost difference as determined by total number of boluses, number of ventilator hours, and length of ICU stay | Throughout the ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Mary B Taylor, M.D., MSCI, Principal Investigator — Vanderbilt University Medical Center Department of Pediatrics Division of Critical Care
Locations (1):
- The Monroe Carell, Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee, United States